CLINICAL TRIAL: NCT00002850
Title: Oral Antibiotic Prophylaxis of Early Infection in Multiple Myeloma
Brief Title: Antibiotic Therapy in Preventing Early Infection in Patients With Multiple Myeloma Who Are Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, UR NCORP Research BAase, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000065093; U10CA037420 (NIH); URCC-U10994 (Other: University of Rochester Cancer Center); NCI-C95-0001 (Other: NIH/NCI DCP); URCC-URRSRB-6993 (Other: University of Rochester IRB); NCI-P96-0073 (Other: NCI); ECOG-U1099 (Other: ECOG)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Infection; Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; infection
MeSH Terms: conditions — Infections; Multiple Myeloma | interventions — Ciprofloxacin; Ofloxacin; Trimethoprim; Sulfamethoxazole; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ciprofloxacin or ofloxacin (Experimental): Quinolone:
  Ciprofloxacin 500 mg every 12 hours or Ofloxacin400 mg every 12 hours.
  Interventions: Drug: ciprofloxacin; Drug: ofloxacin
- TMP-SMX (Experimental): TMP-SMX: 160 mg trimethoprim and 800 mg sulfamethoxazole every 12 hours
  Interventions: Drug: 160 mg trimethoprim and 800 mg sulfamethoxazole
- No prophylaxis (No Intervention): The patient will receive no prophylactic antibiotics.

INTERVENTIONS:
Drug: ciprofloxacin — Begin oral ciprofloxacin when they start chemotherapy for multiple myeloma. Assigned treatment consists of ciprofloxacin (Cipro 500 mg po tablet every 12 hours for two months. The patient will continue to be observed one additional month on study continuing regular myeloma chemotherapy.
  Other Names: Cipro
  Arms: Ciprofloxacin or ofloxacin
Drug: ofloxacin — Begin oral ofloxacin when they start chemotherapy for multiple myeloma. Assigned treatment consists of ofloxacin (500 mg po tablet every 12 hours for two months. The patient will continue to be observed one additional month on study continuing regular myeloma chemotherapy.
  Other Names: Floxin
  Arms: Ciprofloxacin or ofloxacin
Drug: 160 mg trimethoprim and 800 mg sulfamethoxazole — Begin oral TMP-SMX when they start chemotherapy for multiple myeloma. Assigned treatment consists of TMP-SMX (Septra® or Bactrim®) 1 DS tablet [TMP-SMX DS = 160 mg trimethoprim and 800 mg sulfamethoxazole] every 12 hours for two months..
  Other Names: TMP-SMX; Septra; Bactrim
  Arms: TMP-SMX

SUMMARY:
RATIONALE: Giving antibiotics may be effective in preventing or controlling early infection in patients with multiple myeloma and may improve their response to chemotherapy.

PURPOSE: This randomized clinical trial is studying antibiotics to see how well they work compared to no antibiotics in preventing early infection in patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate whether oral antibiotic prophylaxis with co-trimoxazole (TMP-SMX) versus ciprofloxacin (CPFX) or ofloxacin versus no prophylaxis will significantly reduce rates of serious bacterial infections during the first 3 months of chemotherapy in patients with multiple myeloma.
* Determine whether antibiotic prophylaxis with TMP-SMX or CPFX (or ofloxacin) is associated with an increased incidence of nonbacterial infection or an increased rate of infection from organisms resistant to prophylactic antibiotics.
* Evaluate whether oral antibiotic prophylaxis with CPFX or ofloxacin is as effective as TMP-SMX without the associated toxic effects.
* Evaluate whether protection against early infection in multiple myeloma patients can improve their response to initial chemotherapy.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating center. Patients are randomized to 1 of 2treatment arms.

* Arm I: Patients receive co-trimoxazole every 12 hours for 2 months followed by observation for 2 months.
* Arm II: Patients receive oral ciprofloxacin or ofloxacin every 12 hours for 2 months followed by observation for 1 month.
* Arm III: The patient will receive no prophylaxis.

Patients continue their randomly assigned treatment throughout any infection in addition to any treatment needed for infection. Patients also remain on their randomly assigned treatment if chemotherapy is discontinued, changed, or delayed during the 3 month study.

Patients are followed at 6 months, 1 year, and 2 years.

PROJECTED ACCRUAL: A total of 212 patients (71 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion:

* Patient must have a diagnosis of multiple myeloma confirmed by the presence of:
* Bone marrow plasmacytosis with >10% abnormal plasma cells or multiple biopsy-proven plasmacytomas, and at least one of the criteria below must be documented:

  1. Myeloma protein in the serum
  2. Myeloma protein in the urine (free monoclonal light chain)
  3. Radiologic evidence of osteolytic lesions (generalized osteoporosis qualifies only if the bone marrow aspirate contains >20% plasma cells)
* Patients must have no active infection during the prior seven days and be off all antibiotics for the prior seven days.
* Patients cannot have received radiotherapy during the preceding ten days.
* Primary therapy for multiple myeloma must start within three days after entry to this study. For purposes of eligibility for this study, myelosuppressive chemotherapy or high-dose dexamethasone based regimens are acceptable as primary therapy. The high-dose dexamethasone regimen must include, at a minimum, dexamethasone 40 mg per day days 1-4, 9-12, 17-20 for the first cycle and 40 mg per day on days 1-4 of the second cycle.
* Patients who are to receive dexamethasone alone or dexamethasone with thalidomide are among those eligible for this protocol.
* Patients must have a serum creatinine <5.0 mg/dl and not require dialysis at the time of study entry. If patients require dialysis after enrollment, they can continue on the protocol using the adjusted medication guidelines
* Written informed consent must be obtained prior to entry.

Exclusion:

- Patients with smoldering myeloma, history of hypersensitivity to fluoroquinolones or trimethoprim, bone marrow transplant or autologous stem cell rescue planned during the first two months of treatment, patients taking theophylline, or patients previously treated with chemotherapy or high-dose dexamethasone

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 1997-03; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — University of Rochester; Martin M. Oken, MD, Study Chair — CCOP - Metro-Minnesota; Claire Pomeroy, MD, Study Chair — University of California, Davis
Locations (45):
- United States (43):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - CCOP - Northwest, Tacoma, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Pretoria Academic Hospital, Pretoria, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin or Ofloxacin: ciprofloxacin: Begin oral ciprofloxacin when they start chemotherapy for multiple myeloma. Assigned treatment consists of ciprofloxacin (Cipro® 500 mg po tablet every 12 hours for two months. The patient will continue to be observed one additional month on study continuing regular myeloma chemotherapy.
  ofloxacin: Begin oral ofloxacin when they start chemotherapy for multiple myeloma. Assigned treatment consists of ofloxacin (500 mg po tablet every 12 hours for two months. The patient will continue to be observed one additional month on study continuing regular myeloma chemotherapy.
- TMP-SMX: trimethoprim-sulfamethoxazole: Begin oral Trimethoprim-sulfamethoxazole when they start chemotherapy for multiple myeloma. Assigned treatment consists of TMP-SMX (Septra® or Bactrim®) 1 DS tablet [TMP-SMX DS = 160 mg trimethoprim and 800 mg sulfamethoxazole] every 12 hours for two months..
- Observation: Patients observed without intervention and evaluated for SBI for the first 2 months of treatment.
Period: Overall Study
Arm/Group | Ciprofloxacin or Ofloxacin | TMP-SMX | Observation
Started | 69 | 76 | 67
Completed | 64 | 74 | 63
Not Completed | 5 | 2 | 4
Not completed — Death | 4 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients with symptomatic and untreated MM receiving chemotherapy without an active infection during the 7 days prior to initiation of chemotherapy and off antibiotics for the prior 7 days were eligable for this study. They were required to receive myelosuppressive and/or immunosuppressive chemotherapy, and were randomized on a 1:1 basis.
Groups:
- Observation: No prophylaxis: The patient will receive no prophylactic antibiotics.
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin or Ofloxacin | TMP-SMX | Observation | Total
Number analyzed (Participants) | 69 | 76 | 67 | 212
Age, Continuous [Mean (Full Range); unit: years] | 63.7 [32.4 to 86.0] | 62.6 [36.7 to 85.7] | 65.0 [36.7 to 89.3] | 63.2 [32.4 to 89.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 32 | 24 | 79
  Male | 46 | 44 | 43 | 133
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54 | 51 | 55 | 160
  Unknown | 15 | 25 | 12 | 52
Region of Enrollment [Number; unit: participants]
  United States | 69 | 76 | 67 | 212
Infection in last 6 months [Number; unit: participants]
  Yes | 13 | 7 | 8 | 28
  Unknown | 56 | 69 | 59 | 184
Chemotherapy regimen [Number; unit: participants] — VBMCP=vincristine, carmustine, melphalan, cyclophosphamide, and prednisone
  participants
    Melphalan, Prednisone | 11 | 13 | 10 | 34
    VBMCP | 6 | 8 | 8 | 22
    Vincristine, Adriamycin, Dexamethasone | 24 | 17 | 22 | 63
    Other | 28 | 38 | 27 | 93
Eastern Cooperative Oncology Group (ECOG) performance status [Mean (Full Range); unit: units on a scale] — ECOG PERFORMANCE STATUS: Used by doctors and researchers to assess how a patient's disease is progressing.
  0: Fully active, able to carry on pre-disease performance
  1. Restricted in physically strenuous activity but ambulatory; able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on selfcare. Confined to bed or chair
  5. Dead
  units on a scale | 1.0 [0 to 3] | 1.1 [0 to 4] | 0.8 [0 to 4] | 1.0 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing a Serious Bacterial Infection
Description: This study evaluated the impact of prophylactic antibiotics on the incidence of serious bacterial infections (SBIs) during the first 2 months of treatment in patients with newly diagnosed multiple myeloma. Patients with multiple myeloma receiving initial chemotherapy were randomized on a 1:1:1 basis to daily ciprofloxacin, trimethoprim-sulfamethoxazole, or observation and evaluated for SBI for the first 2 months of treatment.
Time Frame: First three months of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ciprofloxacin or Ofloxacin | TMP-SMX | No Prophylaxis
Number analyzed (Participants) | 64 | 74 | 63
percentage of participants | 12.5 [5.6 to 23.2] | 6.8 [2.2 to 15.1] | 15.9 [7.9 to 27.3]
Statistical Analysis 1: Comparison: Ciprofloxacin or Ofloxacin vs TMP-SMX vs No Prophylaxis; H0: There is no significant difference in the incidence of severe bacterial infections among all three arms during the first 2 months of treatment at the two-sided 0.05 significance level. Ha: There is a significant difference in the incidence of severe bacterial infections among all three arms during the first 2 months of treatment at the two-sided 0.05 significance level; Test type: Superiority or Other; p = 0.218, Fisher Exact; Target accrual=70 patients per arm to provide 92% power to detect a difference of 0.31 vs. 0.08 in the proportion of patients with serious infection

ADVERSE EVENTS:
Time Frame: Three months.
Arm/Group | Ciprofloxacin or Ofloxacin | TMP-SMX | Observation
Serious Adverse Events (participants affected / at risk) | 1/69 | 2/76 | 0/67
Other Adverse Events (participants affected / at risk) | 1/69 | 1/76 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin or Ofloxacin (N=69) | TMP-SMX (N=76) | Observation (N=67)
Death (General disorders) | 1 | 0 | 0 — Hospitalized for evaluation of pain, shortness of breath, cough; death
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 — Hospitalized for acute renal failure
Infection, thrush, allergic reaction (Infections and infestations) | 0 | 1 | 0 — Hospitalized for bacterial infection, oral thrush, allergic reaction to sulfa
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin or Ofloxacin (N=69) | TMP-SMX (N=76) | Observation (N=67)
Thrush (Infections and infestations) | 0 | 1 | 0
GI bleed (Gastrointestinal disorders) | 1 | 0 | 0 — Hospitalized with GI bleed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No